CLINICAL TRIAL: NCT06290232
Title: Fetoscopic Laser Photocoagulation in Management of Vasa Previa - FLUMEN Study
Brief Title: Fetoscopic Laser Photocoagulation in Management of Vasa Previa
Acronym: FLUMEN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alireza Shamshirsaz, Chief, Division of Fetal Medicine and Surgery; Director, Maternal Fetal Care Center, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00044498
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Vasa Previa; Pregnancy Complications; Maternal; Procedure; In Utero Procedure Affecting Fetus or Newborn
Keywords: Fetoscope; Fetoscopic Laser Photocoagulation; Low-Lying Fetal Vessels
MeSH Terms: conditions — Vasa Previa; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Fetoscopic Laser Photocoagulation Surgery (Experimental): Pregnant individuals diagnosed with type II vasa previa will undergo fetoscopic laser photocoagulation.
  Interventions: Device: Fetoscopic Laser Photocoagulation

INTERVENTIONS:
Device: Fetoscopic Laser Photocoagulation — Pregnant patients diagnosed with type II vasa previa will undergo fetoscopic laser photocoagulation of the involved fetal vessels. FLP will be performed laparoscopically using a fetoscope (tiny telescope) and a laser device inside of the womb. This procedure will be completed at 30w0d to 32w6d gestational age.
  Other Names: Fetoscopic Laser Ablation

SUMMARY:
In this research study, the investigators want to learn more about the safety and effectiveness of a fetal surgery, known as fetoscopic laser photocoagulation (FLP), for the treatment of a pregnancy condition called vasa previa (VP). Vasa previa is a pregnancy complication that happens when blood vessels from the fetus grow over the entrance to the womb. In a VP pregnancy, natural vaginal birth is deadly for the baby in more than half of cases due to the bursting of VP vessels and severe blood loss. Currently, VP patients are recommended to be closely monitored and often hospitalized once they reach the third trimester of pregnancy. An early delivery by C-section would typically be performed in order to avoid breaking the exposed fetal vessels.

Fetoscopic laser photocoagulation is a minimally invasive surgery in the womb to remove or correct abnormal blood vessels and tissues. In the FLP procedure, the surgeon uses a fetoscope (a tiny telescope) and a laser device to seal off unprotected vessels. While this surgery has been used to treat other pregnancy conditions, it has not yet been proven to be safe and/or effective for the treatment of vasa previa. This treatment aims to eliminate the VP, and, if successful, may have the potential to minimize the risk of bleeding, thereby enabling patients to avoid long hospitalization before delivery. This procedure may enable VP patients to have a vaginal delivery instead of C-section.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patient
* Singleton pregnancy
* Confirmed diagnosis of vasa previa, defined as unprotected fetal vessels running through the membranes at or within 5cm of the internal cervical os. Diagnosis must be confirmed after 26w0d, and before 32w5d
* Able to undergo intervention during 30w0d to 32w6d
* Type II vasa previa in which one placental lobe is considered to be accessory, defined as constituting less than 20% of the total placental mass seen on MRI and US imaging
* Type II vasa previa in which multiple bridging vessels connect the two placental lobes (≥4 vessels), and only 1-2 vessel(s) run through or within 5cm of the internal cervical os
* Patient is eligible to undergo anesthesia
* Patient and biological father of the fetus (if available) are able to provide signed informed consent

Exclusion Criteria:

* Gestational age at referral higher than 32w6d
* Multiple pregnancy
* Vasa previa types I and III
* Type II vasa previa in which the accessory lobe constitutes more than 20% of the total placental mass, as determined by the fetal surgeon during diagnostic fetoscopy
* Type II vasa previa in which all of the bridging vessels between placental lobes are running over the internal cervical os
* Fetal growth restriction, defined as estimated fetal weight or abdominal circumference less than the 10th percentile for gestational age
* Abnormal fetal brain MRI, including delayed maturation, hemorrhage, arterial ischemic injury, abnormal ventricular size, or any congenital anomalies
* Allergy or previous adverse reaction to ancillary medications with no available alternative
* Preterm contractions and PPROM before surgery
* Preeclampsia or uterine anomaly during the current pregnancy
* Placenta previa, low-lying placenta, placenta accreta spectrum disorder
* Suspicion of major recognized congenital syndrome on ultrasound or MRI that is not compatible with postnatal life
* Maternal pre-pregnancy BMI >40
* Active hepatitis B, hepatitis C, or HIV infection
* High risk for congenital fetal bleeding disorders
* Unreliable pregnancy dating due to an irregular menstrual cycle/uncertain last menstrual period with no confirmed dating from first trimester ultrasound
* The surgeon determines that the procedure is not feasible for any other reason after diagnostic fetoscopy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The type of delivery, categorized as vaginal, assisted vaginal, or cesarean section.
Gestational age at delivery | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The duration of pregnancy, measured in completed [weeks + days] from the first day of the last menstrual period (in individuals with regular menses and reliable dating) or determined through first-trimester ultrasound using fetal biometric measurements.
Successful visualization and mapping of vasa previa | When the last (20th) participant undergoes FLP surgery, about 3 years from study start date.
  Confirmation by the performing surgeon that the visualization and mapping of vasa previa by diagnostic fetoscopy matches imaging from US and MRI.
The rate of successful coagulation of the vasa previa - intraoperative imaging | When the last (20th) participant undergoes FLP surgery, about 3 years from study start date.
  Confirmation of the complete coagulation of the vasa previa including the absence of blood flow in involved vessels. This will be measured in the OR directly after FLP surgery by ultrasound.
The rate of successful coagulation of the vasa previa - postoperative imaging | Two weeks after the last (20th) participant undergoes FLP surgery, about 3 years from study start date.
  Confirmation of the complete coagulation of the vasa previa including the absence of blood flow in involved vessels. This will be measured 2 weeks post-surgery by ultrasound and MRI.
The rate of successful coagulation of the vasa previa - pathology | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  Confirmation of the complete coagulation of the vasa previa including the absence of blood flow in involved vessels. This will be measured after delivery during placental analysis by pathology.
Placental function | Two weeks after the last (20th) participant undergoes FLP surgery, about 3 years from study start date.
  Successful maintenance of placental function after surgery. This will be measured by MRI 2 weeks after surgery.

SECONDARY OUTCOMES:
GA at hospital admission | When the last (20th) participant is admitted to the hospital, a little less than 3 years from study start date
  The gestational age at hospital admission before birth.
Duration of hospital stay | When the last (20th) participant is discharged from the hospital, a little more than 3 years from study start date
  The length of hospital stay for the pregnant person will be recorded, from the time of admission to discharge.
Cause for hospital admission | When the last (20th) participant is admitted to the hospital, a little less than 3 years from study start date
  The reason for hospital admission before birth will be recorded.
The rate of spontaneous preterm labor | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The incidence of labor occurring naturally before 37 completed weeks of pregnancy with regular uterine contractions and progressive cervical dilation in the absence of medical or obstetric intervention.
The rate of preterm premature rupture of membranes (PPROM) | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The incidence of PPROM, defined as rupture of the amniotic sac after FLP surgery and before 37 completed weeks of pregnancy.
The rate of placental abruption | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The rate of separation of the placenta from the uterine wall after FLP surgery and before delivery.
The rate of chorioamnionitis | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The rate of infection of the fetal membranes and amniotic fluid after FLP surgery and before delivery.
The rate of chorioamniotic separation | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The rate of separation of the amniotic and chorionic membranes after FLP surgery and before delivery.
Interval from procedure to delivery | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The length of time from FLP surgery to delivery will be recorded in weeks and days.
The rate of fetal growth restriction | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The rate of fetal growth restriction, defined as an estimated fetal weight or abdominal circumference below the 10th percentile for gestational age, at any time after FLP surgery up to delivery.
Fetal brain structure | Two weeks after the last (20th) participant undergoes FLP surgery, about 3 years from study start date
  Normal or abnormal fetal brain structure will be assessed by MRI 2 weeks after surgery.
The rate of NICU admission | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The rate of NICU admission after birth will be recorded
NICU length of stay | When the last baby is discharged from the NICU, a little more than 3 years from study start date
  The number of days that the baby spends in the NICU after birth.
Short term neonatal morbidity | When the last baby is discharged from the hospital, a little more than 3 years from study start date
  The rate of short term morbidity during the first 30 days of life or until hospital discharge, whichever is latest. Short-term morbidity includes neurological problems, gastrointestinal problems, respiratory problems, infections, and other problems associated with prematurity including but not limited to: necrotizing enterocolitis, bronchopulmonary dysplasia, respiratory distress syndrome, neonatal sepsis, neonatal intensive care unit admission and need for extracorporeal membrane oxygenation (ECMO).
Neonatal survival | When the last baby is discharged from the hospital, a little more than 3 years from study start date
  The rate of neonates surviving to 30 days of age, or hospital discharge, whichever is latest.
Maternal mental health score | Two weeks after the last (20th) participant undergoes FLP surgery, about 3 years from study start date
  The Postpartum Depression Screening Scale (PDSS) - Antenatal Version will be used to assess and compare the levels of depression and anxiety before and after FLP surgery. This assessment will be given once before surgery, and once again 4-8 weeks later (at least 2 weeks after surgery).
Postnatal examination of the placenta | When the last (20th) participant reaches delivery, a little more than 3 years from study start date
  The placenta will be examined for disrupted or ruptured vessels after dye staining. Secondary changes in the accessory lobe will also be checked, which are features resulting from cessation of blood supply due to prior ablation. These could include fibrin deposition, evidence of hypoxia in the chorionic villi, eventual necrosis, and parenchymal atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Shamshirsaz, MD, Principal Investigator — Director, Maternal Fetal Care Center; Chief, Division of Fetal Medicine and Surgery
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oyelese KO, Turner M, Lees C, Campbell S. Vasa previa: an avoidable obstetric tragedy. Obstet Gynecol Surv. 1999 Feb;54(2):138-45. doi: 10.1097/00006254-199902000-00024. PMID 9950006
- [Background] Pavalagantharajah S, Villani LA, D'Souza R. Vasa previa and associated risk factors: a systematic review and meta-analysis. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100117. doi: 10.1016/j.ajogmf.2020.100117. Epub 2020 Apr 15. PMID 33345868
- [Background] Zhang W, Giacchino T, Chanyarungrojn PA, Ionescu O, Akolekar R. Incidence of vasa praevia: a systematic review and meta-analysis. BMJ Open. 2023 Sep 20;13(9):e075245. doi: 10.1136/bmjopen-2023-075245. PMID 37730391
- [Background] Oyelese Y, Chavez MR, Yeo L, Giannina G, Kontopoulos EV, Smulian JC, Scorza WE. Three-dimensional sonographic diagnosis of vasa previa. Ultrasound Obstet Gynecol. 2004 Aug;24(2):211-5. doi: 10.1002/uog.1097. No abstract available. PMID 15287065
- [Background] Silver RM. Vasa praevia: improved diagnosis through recognition of risk factors. BJOG. 2016 Jul;123(8):1288. doi: 10.1111/1471-0528.13870. Epub 2016 Feb 5. No abstract available. PMID 26846196
- [Background] Oyelese Y, Smulian JC. Placenta previa, placenta accreta, and vasa previa. Obstet Gynecol. 2006 Apr;107(4):927-41. doi: 10.1097/01.AOG.0000207559.15715.98. PMID 16582134
- [Background] Zhang W, Geris S, Al-Emara N, Ramadan G, Sotiriadis A, Akolekar R. Perinatal outcome of pregnancies with prenatal diagnosis of vasa previa: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2021 May;57(5):710-719. doi: 10.1002/uog.22166. PMID 32735754
- [Background] Ranzini AC, Oyelese Y. How to screen for vasa previa. Ultrasound Obstet Gynecol. 2021 May;57(5):720-725. doi: 10.1002/uog.23520. No abstract available. PMID 33085148
- [Background] Oyelese Y. Re: Incidence of and risk factors for vasa praevia: a systematic review: Vasa praevia screening. BJOG. 2017 Jan;124(1):162. doi: 10.1111/1471-0528.14013. No abstract available. PMID 28009122
- [Background] Society of Maternal-Fetal (SMFM) Publications Committee; Sinkey RG, Odibo AO, Dashe JS. #37: Diagnosis and management of vasa previa. Am J Obstet Gynecol. 2015 Nov;213(5):615-9. doi: 10.1016/j.ajog.2015.08.031. Epub 2015 Aug 18. PMID 26292048
- [Background] Jain V, Gagnon R. Guideline No. 439: Diagnosis and Management of Vasa Previa. J Obstet Gynaecol Can. 2023 Jul;45(7):506-518. doi: 10.1016/j.jogc.2023.05.009. Epub 2023 May 18. PMID 37209787
- [Background] Oyelese Y. Prenatally Diagnosed Vasa Previa: A Single-Institution Series of 96 Cases. Obstet Gynecol. 2017 Mar;129(3):581-582. doi: 10.1097/AOG.0000000000001919. No abstract available. PMID 28225412
- [Background] Klahr R, Fox NS, Zafman K, Hill MB, Connolly CT, Rebarber A. Frequency of spontaneous resolution of vasa previa with advancing gestational age. Am J Obstet Gynecol. 2019 Dec;221(6):646.e1-646.e7. doi: 10.1016/j.ajog.2019.06.040. Epub 2019 Jun 21. PMID 31233708
- [Background] Bronsteen R, Whitten A, Balasubramanian M, Lee W, Lorenz R, Redman M, Goncalves L, Seubert D, Bauer S, Comstock C. Vasa previa: clinical presentations, outcomes, and implications for management. Obstet Gynecol. 2013 Aug;122(2 Pt 1):352-357. doi: 10.1097/AOG.0b013e31829cac58. PMID 23969805
- [Background] Westcott JM, Simpson S, Chasen S, Vieira L, Stone J, Doulaveris G, Dar P, Bernstein PS, Atallah F, Dolin CD, Roman AS. Prenatally diagnosed vasa previa: association with adverse obstetrical and neonatal outcomes. Am J Obstet Gynecol MFM. 2020 Nov;2(4):100206. doi: 10.1016/j.ajogmf.2020.100206. Epub 2020 Aug 15. PMID 33345921
- [Background] Chmait RH, Chavira E, Kontopoulos EV, Quintero RA. Third trimester fetoscopic laser ablation of type II vasa previa. J Matern Fetal Neonatal Med. 2010 May;23(5):459-62. doi: 10.1080/14767050903156718. PMID 19637106
- [Background] Erfani H, Haeri S, Shainker SA, Saad AF, Ruano R, Dunn TN, Rezaei A, Aalipour S, Nassr AA, Shamshirsaz AA, Vaughn M, Lindsley W, Spiel MH, Shazly SA, Ibirogba ER, Clark SL, Saade GR, Belfort MA, Shamshirsaz AA. Vasa previa: a multicenter retrospective cohort study. Am J Obstet Gynecol. 2019 Dec;221(6):644.e1-644.e5. doi: 10.1016/j.ajog.2019.06.006. Epub 2019 Jun 13. PMID 31201807
- [Background] Sutera M, Garofalo A, Pilloni E, Parisi S, Alemanno MG, Menato G, Sciarrone A, Viora E. Vasa previa: when antenatal diagnosis can change fetal prognosis. J Perinat Med. 2021 May 4;49(7):915-922. doi: 10.1515/jpm-2020-0559. Print 2021 Sep 27. PMID 33939903
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Burton GJ, Collins SL, Silver R; Royal College of Obstetricians and Gynaecologists. Vasa Praevia: Diagnosis and Management: Green-top Guideline No. 27b. BJOG. 2019 Jan;126(1):e49-e61. doi: 10.1111/1471-0528.15307. Epub 2018 Sep 27. No abstract available. PMID 30260094
- [Background] Green A, Chiu S, Manor E, Smith L, Oyelese Y. The association of gestational age at delivery with neonatal outcomes in prenatally diagnosed vasa previa. J Matern Fetal Neonatal Med. 2022 Dec;35(25):10162-10167. doi: 10.1080/14767058.2022.2122040. Epub 2022 Sep 11. PMID 36093853
- [Background] Swank ML, Garite TJ, Maurel K, Das A, Perlow JH, Combs CA, Fishman S, Vanderhoeven J, Nageotte M, Bush M, Lewis D; Obstetrix Collaborative Research Network. Vasa previa: diagnosis and management. Am J Obstet Gynecol. 2016 Aug;215(2):223.e1-6. doi: 10.1016/j.ajog.2016.02.044. Epub 2016 Mar 2. PMID 26944186
- [Background] Catanzarite V, Cousins L, Daneshmand S, Schwendemann W, Casele H, Adamczak J, Tith T, Patel A. Prenatally Diagnosed Vasa Previa: A Single-Institution Series of 96 Cases. Obstet Gynecol. 2016 Nov;128(5):1153-1161. doi: 10.1097/AOG.0000000000001680. PMID 27741189
- [Background] Mitchell SJ, Ngo G, Maurel KA, Hasegawa J, Arakaki T, Melcer Y, Maymon R, Vendittelli F, Shamshirsaz AA, Erfani H, Shainker SA, Saad AF, Treadwell MC, Roman AS, Stone JL, Rolnik DL. Timing of birth and adverse pregnancy outcomes in cases of prenatally diagnosed vasa previa: a systematic review and meta-analysis. Am J Obstet Gynecol. 2022 Aug;227(2):173-181.e24. doi: 10.1016/j.ajog.2022.03.006. Epub 2022 Mar 10. PMID 35283090
- [Background] Oyelese Y, Iammatteo M, Domnitz S, Chavez MR. Vasa previa: avoiding incising the membranes at cesarean delivery. Am J Obstet Gynecol. 2022 Nov;227(5):770-772. doi: 10.1016/j.ajog.2022.07.010. Epub 2022 Jul 15. PMID 35843270
- [Background] Oyelese Y, Javinani A, Shamshirsaz AA. Vasa Previa. Obstet Gynecol. 2023 Sep 1;142(3):503-518. doi: 10.1097/AOG.0000000000005287. Epub 2023 Aug 3. PMID 37590981
- [Background] Monson MA, Chmait RH, Einerson B. Fetoscopic Laser Ablation of Type II Vasa Previa: A Cost Benefit Analysis. Am J Perinatol. 2024 May;41(S 01):e2454-e2462. doi: 10.1055/s-0043-1771262. Epub 2023 Jul 21. PMID 37494587
- [Background] Ibirogba ER, Shazly SA, Chmait RH, Ruano R. Is there a role for fetoscopic laser ablation therapy in Type-2 vasa previa? Ultrasound Obstet Gynecol. 2019 Nov;54(5):696. doi: 10.1002/uog.20251. No abstract available. PMID 30801796
- [Background] Quintero RA, Kontopoulos EV, Bornick PW, Allen MH. In utero laser treatment of type II vasa previa. J Matern Fetal Neonatal Med. 2007 Dec;20(12):847-51. doi: 10.1080/14767050701731605. PMID 18050017
- [Background] Chmait RH, Catanzarite V, Chon AH, Korst LM, Llanes A, Ouzounian JG. Fetoscopic Laser Ablation Therapy for Type II Vasa Previa. Fetal Diagn Ther. 2020;47(9):682-688. doi: 10.1159/000508044. Epub 2020 Jul 6. PMID 32629451
- [Background] Papanna R, Agarwal N, Bergh EP, Brock C, Espinoza J, Johnson A. Fetoscopic laser ablation in pregnancies with Type-II vasa previa. Ultrasound Obstet Gynecol. 2023 Jun;61(6):779-781. doi: 10.1002/uog.26153. No abstract available. PMID 36609872
- [Background] Hosseinzadeh P, Shamshirsaz AA, Cass DL, Espinoza J, Lee W, Salmanian B, Ruano R, Belfort MA. Fetoscopic laser ablation of vasa previa in pregnancy complicated by giant fetal cervical lymphatic malformation. Ultrasound Obstet Gynecol. 2015 Oct;46(4):507-8. doi: 10.1002/uog.14796. No abstract available. PMID 25612246
- [Background] Noble KG, Fifer WP, Rauh VA, Nomura Y, Andrews HF. Academic achievement varies with gestational age among children born at term. Pediatrics. 2012 Aug;130(2):e257-64. doi: 10.1542/peds.2011-2157. Epub 2012 Jul 2. PMID 22753563
- [Background] Sorensen A, Sinding M, Peters DA, Petersen A, Frokjaer JB, Christiansen OB, Uldbjerg N. Placental oxygen transport estimated by the hyperoxic placental BOLD MRI response. Physiol Rep. 2015 Oct;3(10):e12582. doi: 10.14814/phy2.12582. PMID 26471757
- [Background] Luo J, Abaci Turk E, Bibbo C, Gagoski B, Roberts DJ, Vangel M, Tempany-Afdhal CM, Barnewolt C, Estroff J, Palanisamy A, Barth WH, Zera C, Malpica N, Golland P, Adalsteinsson E, Robinson JN, Grant PE. In Vivo Quantification of Placental Insufficiency by BOLD MRI: A Human Study. Sci Rep. 2017 Jun 16;7(1):3713. doi: 10.1038/s41598-017-03450-0. PMID 28623277
- [Background] Schabel MC, Roberts VHJ, Gibbins KJ, Rincon M, Gaffney JE, Streblow AD, Wright AM, Lo JO, Park B, Kroenke CD, Szczotka K, Blue NR, Page JM, Harvey K, Varner MW, Silver RM, Frias AE. Quantitative longitudinal T2* mapping for assessing placental function and association with adverse pregnancy outcomes across gestation. PLoS One. 2022 Jul 19;17(7):e0270360. doi: 10.1371/journal.pone.0270360. eCollection 2022. PMID 35853003
- [Background] Sinding M, Sorensen A, Hansen DN, Peters DA, Frokjaer JB, Petersen AC. T2* weighted placental MRI in relation to placental histology and birth weight. Placenta. 2021 Oct;114:52-55. doi: 10.1016/j.placenta.2021.07.304. Epub 2021 Aug 24. PMID 34461455
- [Background] Sorensen A, Peters D, Frund E, Lingman G, Christiansen O, Uldbjerg N. Changes in human placental oxygenation during maternal hyperoxia estimated by blood oxygen level-dependent magnetic resonance imaging (BOLD MRI). Ultrasound Obstet Gynecol. 2013 Sep;42(3):310-4. doi: 10.1002/uog.12395. PMID 23303592
- [Background] Huen I, Morris DM, Wright C, Parker GJ, Sibley CP, Johnstone ED, Naish JH. R1 and R2 * changes in the human placenta in response to maternal oxygen challenge. Magn Reson Med. 2013 Nov;70(5):1427-33. doi: 10.1002/mrm.24581. Epub 2012 Dec 27. PMID 23280967
- [Background] Abaci Turk E, Abulnaga SM, Luo J, Stout JN, Feldman HA, Turk A, Gagoski B, Wald LL, Adalsteinsson E, Roberts DJ, Bibbo C, Robinson JN, Golland P, Grant PE, Barth WH Jr. Placental MRI: Effect of maternal position and uterine contractions on placental BOLD MRI measurements. Placenta. 2020 Jun;95:69-77. doi: 10.1016/j.placenta.2020.04.008. Epub 2020 Apr 22. PMID 32452404
- [Background] Abaci Turk E, Stout JN, Feldman HA, Gagoski B, Zhou C, Tamen R, Manhard MK, Adalsteinsson E, Roberts DJ, Golland P, Grant PE, Barth WH Jr. Change in T2* measurements of placenta and fetal organs during Braxton Hicks contractions. Placenta. 2022 Oct;128:69-71. doi: 10.1016/j.placenta.2022.08.011. Epub 2022 Aug 29. PMID 36087451
- [Background] Vasung L, Xu J, Abaci-Turk E, Zhou C, Holland E, Barth WH, Barnewolt C, Connolly S, Estroff J, Golland P, Feldman HA, Adalsteinsson E, Grant PE. Cross-Sectional Observational Study of Typical in utero Fetal Movements Using Machine Learning. Dev Neurosci. 2023;45(3):105-114. doi: 10.1159/000528757. Epub 2022 Dec 20. PMID 36538911
- [Background] Abaci Turk E, Yun HJ, Feldman HA, Lee JY, Lee HJ, Bibbo C, Zhou C, Tamen R, Grant PE, Im K. Association between placental oxygen transport and fetal brain cortical development: a study in monochorionic diamniotic twins. Cereb Cortex. 2024 Jan 14;34(1):bhad383. doi: 10.1093/cercor/bhad383. PMID 37885155
- [Background] Stout JN, Liao C, Gagoski B, Turk EA, Feldman HA, Bibbo C, Barth WH Jr, Shainker SA, Wald LL, Grant PE, Adalsteinsson E. Quantitative T1 and T2 mapping by magnetic resonance fingerprinting (MRF) of the placenta before and after maternal hyperoxia. Placenta. 2021 Oct;114:124-132. doi: 10.1016/j.placenta.2021.08.058. Epub 2021 Aug 24. PMID 34537569
- [Background] Fetal Growth Restriction: ACOG Practice Bulletin, Number 227. Obstet Gynecol. 2021 Feb 1;137(2):e16-e28. doi: 10.1097/AOG.0000000000004251. PMID 33481528
- [Background] Langer O, Sonnendecker EW. Characteristics and management of intrapartum prolonged fetal bradycardia. Br J Obstet Gynaecol. 1982 Nov;89(11):904-12. doi: 10.1111/j.1471-0528.1982.tb05055.x. PMID 7171497
- [Background] Thurlow JA, Kinsella SM. Intrauterine resuscitation: active management of fetal distress. Int J Obstet Anesth. 2002 Apr;11(2):105-16. doi: 10.1054/ijoa.2001.0933. PMID 15321562
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Martins JG, Biggio JR, Abuhamad A. Society for Maternal-Fetal Medicine Consult Series #52: Diagnosis and management of fetal growth restriction: (Replaces Clinical Guideline Number 3, April 2012). Am J Obstet Gynecol. 2020 Oct;223(4):B2-B17. doi: 10.1016/j.ajog.2020.05.010. Epub 2020 May 12. PMID 32407785
- [Background] Beck CT, Gable RK. Postpartum Depression Screening Scale: development and psychometric testing. Nurs Res. 2000 Sep-Oct;49(5):272-82. doi: 10.1097/00006199-200009000-00006. PMID 11009122
- [Background] Beck CT, Gable RK. Further validation of the Postpartum Depression Screening Scale. Nurs Res. 2001 May-Jun;50(3):155-64. doi: 10.1097/00006199-200105000-00005. PMID 11393637
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 171: Management of Preterm Labor. Obstet Gynecol. 2016 Oct;128(4):e155-64. doi: 10.1097/AOG.0000000000001711. PMID 27661654
- [Background] Chmait RH, Kontopoulos EV, Chon AH, Korst LM, Llanes A, Quintero RA. Amniopatch treatment of iatrogenic preterm premature rupture of membranes (iPPROM) after fetoscopic laser surgery for twin-twin transfusion syndrome. J Matern Fetal Neonatal Med. 2017 Jun;30(11):1349-1354. doi: 10.1080/14767058.2016.1214123. Epub 2016 Aug 10. PMID 27686840
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Tita AT, Andrews WW. Diagnosis and management of clinical chorioamnionitis. Clin Perinatol. 2010 Jun;37(2):339-54. doi: 10.1016/j.clp.2010.02.003. PMID 20569811
- [Background] Nassr AA, Hessami K, Shazly SA, Meshinchi N, Corroenne R, Espinoza J, Donepudi R, Sanz Cortes M, Belfort MA, Shamshirsaz AA. Perinatal outcomes of iatrogenic chorioamniotic separation following fetoscopic surgery: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2021 Sep;58(3):347-353. doi: 10.1002/uog.23588. PMID 33428299
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069
- [Background] D'Souza R, Villani L, Hall C, Seyoum M, Kingdom J, Krznaric M, Donnolley N, Javid N. Core outcome set for studies on pregnant women with vasa previa (COVasP): a study protocol. BMJ Open. 2020 Jul 19;10(7):e034018. doi: 10.1136/bmjopen-2019-034018. PMID 32690497
- [Background] Sacco A, Van der Veeken L, Bagshaw E, Ferguson C, Van Mieghem T, David AL, Deprest J. Maternal complications following open and fetoscopic fetal surgery: A systematic review and meta-analysis. Prenat Diagn. 2019 Mar;39(4):251-268. doi: 10.1002/pd.5421. Epub 2019 Feb 27. PMID 30703262